CLINICAL TRIAL: NCT03303079
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial Evaluating the Efficacy and Safety of Subcutaneous Administration of TEV-48125 for the Preventive Treatment of Chronic Migraine
Brief Title: Efficacy and Safety of Subcutaneous Administration of TEV-48125 for the Preventive Treatment of Chronic Migraine
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 406-102-00001; JapicCTI-173723 (Other: Japic)
Record Dates: First submitted 2017-10-02; First posted 2017-10-05 (Actual); Results first posted 2021-06-15 (Actual); Last update posted 2021-06-15 (Actual); Status verified 2021-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — fremanezumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TEV-48125 (675/225/225 mg) group (Experimental): TEV-48125 will be subcutaneously administered once monthly for 3 months (675/225/225 mg).
  Interventions: Drug: TEV-48125
- TEV-48125 (675 mg/placebo/placebo) group (Experimental): TEV-48125 or placebo will be subcutaneously administered once monthly for 3 months (675 mg/ placebo/placebo).
  Interventions: Drug: TEV-48125 or placebo
- Placebo group (Placebo Comparator): Placebo will be subcutaneously administered once monthly for 3 months (placebo/placebo/placebo).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TEV-48125 — TEV-48125 will be subcutaneously administered once monthly for 3 months.
  Arms: TEV-48125 (675/225/225 mg) group
Drug: TEV-48125 or placebo — TEV-48125 or placebo will be subcutaneously administered once monthly for 3 months.
  Arms: TEV-48125 (675 mg/placebo/placebo) group
Drug: Placebo — Placebo will be subcutaneously administered once monthly for 3 months.
  Arms: Placebo group

SUMMARY:
To evaluate the efficacy and safety of subcutaneous (SC) administration of TEV-48125 [monthly TEV-48125 225 mg (loading dose only: 675 mg) and TEV-48125 675 mg once over a period of 3 months] compared with placebo for preventive treatment in Chronic Migraine patients

ELIGIBILITY:
Inclusion Criteria:

* Patient has a history of migraine (according to The International Classification of Headache Disorders, third edition [beta version] criteria) or clinical judgment suggests a migraine diagnosis
* Patient fulfills the criteria for Chronic migraine in baseline information collected during the 28 day screening period
* Not using preventive migraine medications for migraine or other medical conditions or using no more than 1 preventive migraine medication for migraine or other medical conditions if the dose and regimen have been stable for at least 2 months prior to giving informed consent.
* Patient demonstrates compliance with the electronic headache diary during the screening period by entry of headache data on a minimum of 24 of 28 days and the entered data is judged appropriate by the investigator.

Exclusion Criteria:

* Patients who have previously failed (lack of efficacy) 2 or more of the clusters of the medications for treatment of migraine after use for at least 3 months at accepted migraine therapeutic doses
* Patient suffers from unremitting headaches, defined as having headaches for more than 80% of the time that he/she is awake, and less than 4 days without headache per month. Daily headache is acceptable if the patient has headaches 80% or less of the time they are awake on most days.
* Hematological, cardiac, renal, endocrine, pulmonary, gastrointestinal, genitourinary, neurologic, hepatic, or ocular disease considered clinically significant in the judgment of the investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 571 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2019-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Saitama Medical University Hospital, Iruma, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Takeshima T, Nakai M, Shibasaki Y, Ishida M, Kim BK, Ning X, Koga N. Early onset of efficacy with fremanezumab in patients with episodic and chronic migraine: subanalysis of two phase 2b/3 trials in Japanese and Korean patients. J Headache Pain. 2022 Feb 9;23(1):24. doi: 10.1186/s10194-022-01393-0. PMID 35139816

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TEV-48125 (675/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Started | 189 | 191 | 191
Completed | 182 | 180 | 179
Not Completed | 7 | 11 | 12
Not completed — Adverse Event | 0 | 1 | 3
Not completed — Protocol Violation | 5 | 4 | 7
Not completed — Withdrawal by Subject | 2 | 4 | 2
Not completed — Other than specified | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TEV-48125 (675/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group | Total
Number analyzed (Participants) | 189 | 191 | 191 | 571
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 187 | 184 | 190 | 561
  >=65 years | 2 | 7 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (10.2) | 43.5 (10.2) | 42.1 (10.2) | 42.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 165 | 163 | 491
  Male | 26 | 26 | 28 | 80
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 189 | 191 | 191 | 571
Region of Enrollment [Number; unit: participants]
  Japan | 159 | 159 | 161 | 479
  South Korea | 30 | 32 | 30 | 92

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in the Monthly (28 Day) Average Number of Headache Days of at Least Moderate Severity During the 12-week Period After the First Dose of Investigational Medicinal Product (IMP)
Description: Headache-related efficacy endpoints were derived from headache variables collected using an eDiary. On each day, subjects entered headache data in the electronic headache diary for the previous 24-hour period. Subjects who had experienced headache on the previous day answered questions about the headache (ie, occurrence of headache, duration of headache, maximum severity of headache, presence/absence of associated symptoms, and use of acute headache medications). Overall headache duration was recorded numerically, in hours, as well as number of hours with headache of at least moderate severity. If headache was reported, then headache severity was subjectively rated by the subject as mild, moderate, or severe.
  Subjects also recorded the presence or absence of photophobia, phonophobia, nausea, or vomiting, and the status of use of any acute headache medications.
Time Frame: Baseline, 12 weeks
Population: Full Analysis set (FAS): Subjects who received the IMP at least once and had baseline and Week 12 data on monthly average number of headache days of at least moderate severity
Measure: Mean (Standard Error); unit: days/month
Arm/Group | TEV-48125 (675/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 187 | 189 | 190
days/month | -4.12 (0.43) | -4.14 (0.43) | -2.45 (0.43)

2. Secondary Outcome: Mean Change From Baseline in the Monthly Average Number of Migraine Days During the 12-week Period After the First Dose of IMP
Description: as for outcome 1
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days/month
Arm/Group | TEV-48125 (675/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 187 | 189 | 190
days/month | -4.90 (0.50) | -4.07 (0.49) | -2.79 (0.49)

3. Secondary Outcome: Proportion of Subjects Reaching at Least 50% Reduction in the Monthly Average Number of Headache Days of at Least Moderate Severity During the 12-week Period After the First Dose of IMP
Description: as for outcome 1
Time Frame: 12 weeks
Population: Full Analysis set (FAS): Subjects who received the IMP at least once and had baseline and Week 12 data on monthly average number of headache days of at least moderate severity "Overall Number of Participants Analyzed" = the number of subjects meeting responder criteria
Measure: Number; unit: percentage of participants
Arm/Group | TEV-48125 (675/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 54 | 55 | 25
percentage of participants | 29.0 | 29.1 | 13.2

4. Secondary Outcome: Mean Change From Baseline in the Monthly Average Number of Days With Use of Any Acute Headache Medications During the 12-week Period After the First Dose of IMP
Description: Headache-related efficacy endpoints were derived from headache variables collected using an eDiary. On each day, subjects entered headache data in the electronic headache diary for the previous 24-hour period. Subjects who had experienced headache on the previous day answered questions about the headache (ie, occurrence of headache, duration of headache, maximum severity of headache, presence/absence of associated symptoms, and use of acute headache medications).
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days/month
Arm/Group | TEV-48125 (675/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 187 | 189 | 190
days/month | -3.74 (0.44) | -3.87 (0.43) | -2.44 (0.43)

5. Secondary Outcome: Mean Change From Baseline in the Monthly Average Number of Headache Days of at Least Moderate Severity During the 12-week Period After the First Dose of IMP in Subjects Not Receiving Concomitant Preventive Migraine Medications
Description: Headache-related efficacy endpoints were derived from headache variables collected using an eDiary. On each day, subjects entered headache data in the electronic headache diary for the previous 24-hour period. Subjects who had experienced headache on the previous day answered questions about the headache (ie, occurrence of headache, duration of headache, maximum severity of headache, presence/absence of associated symptoms, and use of acute headache medications). Overall headache duration was recorded numerically, in hours, as well as number of hours with headache of at least moderate severity. If headache was reported, then headache severity was subjectively rated by the subject as mild, moderate, or severe.
  Subjects also recorded the presence or absence of photophobia, phonophobia, nausea, or vomiting, and the status of use of any acute headache medications."
Time Frame: Baseline, 12 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: days/month
Arm/Group | TEV-48125 (675/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 149 | 149 | 149
days/month | -3.74 (0.44) | -3.87 (0.43) | -2.44 (0.43)

6. Secondary Outcome: Mean Change From Baseline in Disability Score, as Measured by 6-Item Headache Impact Test (HIT-6) at 4 Weeks After the Final (Third) Dose of IMP
Description: Subjects assessed the impact of headache on social functioning, role functioning, vitality, cognitive functioning, and psychological distress, using the HIT-6. The HIT-6 total score will be obtained from summation of the 6 question points.Each question is answered on the scale ranging with the following response options: 6 points (never), 8 points (rarely), 10 points (sometimes), 11 points (very often), and 13 points (always).
Time Frame: Baseline, 4 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | TEV-48125 (675/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
Number analyzed (Participants) | 182 | 180 | 179
score on a scale | -8.06 (0.70) | -8.03 (0.68) | -6.49 (0.68)

ADVERSE EVENTS:
Time Frame: Double-blind treatment period (12 weeks)
Description: Safety set (SS):Subjects who received the IMP at least once
Arm/Group | TEV-48125 (675/225/225 mg) Group | TEV-48125 (675 mg/Placebo/Placebo) Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/188 | 0/190 | 0/191
Serious Adverse Events (participants affected / at risk) | 3/188 | 1/190 | 1/191
Other Adverse Events (participants affected / at risk) | 115/188 | 116/190 | 117/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEV-48125 (675/225/225 mg) Group (N=188) | TEV-48125 (675 mg/Placebo/Placebo) Group (N=190) | Placebo Group (N=191)
Brain contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TEV-48125 (675/225/225 mg) Group (N=188) | TEV-48125 (675 mg/Placebo/Placebo) Group (N=190) | Placebo Group (N=191)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 2
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1
Palpitations (Cardiac disorders) | 2 | 0 | 1
Prinzmetal angina (Cardiac disorders) | 1 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 1
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 0
Deafness neurosensory (Ear and labyrinth disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 0 | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1 | 0
Dry eye (Eye disorders) | 2 | 0 | 0
Astigmatism (Eye disorders) | 1 | 0 | 0
Conjunctival cyst (Eye disorders) | 1 | 0 | 0
Conjunctivitis allergic (Eye disorders) | 1 | 0 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0
Asthenopia (Eye disorders) | 0 | 1 | 0
Blepharospasm (Eye disorders) | 0 | 0 | 1
Chalazion (Eye disorders) | 0 | 0 | 1
Retinopathy solar (Eye disorders) | 0 | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 3 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3 | 2
Nausea (Gastrointestinal disorders) | 2 | 5 | 2
Tooth loss (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 2 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 0 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 0 | 1
Lumbar hernia (Gastrointestinal disorders) | 0 | 1 | 0
Periodontal inflammation (Gastrointestinal disorders) | 0 | 1 | 0
Salivary gland mass (Gastrointestinal disorders) | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0
Injection site induration (General disorders) | 33 | 23 | 24
Injection site erythema (General disorders) | 29 | 23 | 21
Injection site pain (General disorders) | 14 | 24 | 17
Injection site pruritus (General disorders) | 10 | 3 | 5
Injection site swelling (General disorders) | 3 | 2 | 0
Injection site haemorrhage (General disorders) | 1 | 3 | 0
Injection site rash (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 1 | 2
Chest pain (General disorders) | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 1 | 0
Injection site bruising (General disorders) | 0 | 0 | 2
Injection site dermatitis (General disorders) | 0 | 1 | 0
Injection site inflammation (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Thirst (General disorders) | 0 | 1 | 0
Seasonal allergy (Immune system disorders) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 30 | 40 | 36
Influenza (Infections and infestations) | 4 | 1 | 3
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 0
Gastroenteritis (Infections and infestations) | 2 | 3 | 1
Herpes virus infection (Infections and infestations) | 2 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 2 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Gingivitis (Infections and infestations) | 1 | 1 | 2
Kaposi's varicelliform eruption (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 1 | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 1
Vulvitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 4 | 1
Helicobacter infection (Infections and infestations) | 0 | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 0 | 1
Hordeolum (Infections and infestations) | 0 | 1 | 1
Parotitis (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Pulpitis dental (Infections and infestations) | 0 | 0 | 1
Streptococcal infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Stab wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dental restoration failure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 2 | 0
Muscle contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post-traumatic neck syndrome (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Urine leukocyte esterase positive (Investigations) | 2 | 1 | 0
Weight decreased (Investigations) | 2 | 2 | 2
Alanine aminotransferase increased (Investigations) | 1 | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 2 | 0
Blood glucose increased (Investigations) | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 1 | 0
Blood pressure increased (Investigations) | 0 | 2 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 1
Weight increased (Investigations) | 0 | 1 | 1
White blood cell count increased (Investigations) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Decreased appetite (Investigations) | 0 | 0 | 1
Diabetic complication (Metabolism and nutrition disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spinal deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 3 | 2 | 3
Headache (Nervous system disorders) | 3 | 1 | 1
Syncope (Nervous system disorders) | 2 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0
Hypersomnia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 1 | 3 | 2
Monoplegia (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Presyncope (Nervous system disorders) | 1 | 0 | 0
Amnestic disorder (Nervous system disorders) | 0 | 0 | 1
Dizziness postural (Nervous system disorders) | 0 | 1 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 2
Depression (Psychiatric disorders) | 2 | 0 | 0
Alcoholic hangover (Psychiatric disorders) | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Mental fatigue (Psychiatric disorders) | 0 | 0 | 1
Panic disorder (Psychiatric disorders) | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Premenstrual syndrome (Reproductive system and breast disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Reflux laryngitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 2 | 1 | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 | 0 | 2
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Solar dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Peripheral coldness (Vascular disorders) | 1 | 0 | 0
Neurogenic shock (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT03303079/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT03303079/SAP_001.pdf